CLINICAL TRIAL: NCT02473588
Title: Comparison of Retia Medical (Long Time Interval Analysis) to Deltex Esophageal Doppler for Cardiac Output Measurement
Brief Title: Long Time Interval Analysis for Non Invasive Measurement of Cardiac Output
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robert Thiele, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18022
Record Dates: First submitted 2015-06-11; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LTIA Group (Other): Patients in the LTIA Group (all patients) will have blood pressure recorded continuously. LTIA will be used to measure stroke volume and cardiac output after the completion of data collection
  Interventions: Device: Retia Medical Long Time Interval Analysis

INTERVENTIONS:
Device: Retia Medical Long Time Interval Analysis — Retia Medical "Long Time Interval Analysis" will be used to analyze the blood pressure tracing of patients having surgery who have an arterial catheter

SUMMARY:
A group of engineers at Michigan State developed a novel waveform analysis technique ("Long Time Interval Analysis" [LTIA]) that attempts to estimate cardiac output non-invasively. Retrospective comparison of LTIA to invasive techniques (e.g. thermodilution) suggest acceptable agreement. Thus, a prospective trial of LTIA is warranted. This study compares LTIA to a validated measure of cardiac output - esophageal Doppler monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Undergoing hepatobiliary surgery (open or laparoscopic) requiring general anesthesia as part of the patient's clinical care
* Attending anesthesiologist plans to place an intra-arterial catheter for routine care
* Attending anesthesiologist believes that non-invasive cardiac output monitoring would benefit the patient

Exclusion Criteria:

* Minors (17 years or younger)
* Parturient (pregnant women)
* Cognitively impaired
* Unable to sign informed consent form
* Prisoner
* Prior esophageal surgery
* Moderate to severe aortic regurgitation
* Mechanical cardiac support (e.g., intra-aortic balloon pump)
* Severe, persistent arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pearson Correlation Coefficient | Data collected in first 20 minutes of anesthesia/surgery will be recorded; Pearson correlation coefficient will be calculated after all 60 subjects have been enrolled
  Correlation between change in CO from LTIA vs. change in CO from esophageal Doppler

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States